CLINICAL TRIAL: NCT01890902
Title: A Randomized, Multicenter, Double-Blind, Parallel-Group Study to Assess the Efficacy and Safety of Impracor (Ketoprofen 10% Cream) Compared With Placebo in the Treatment of Acute Pain (Flare) Associated With Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of Impracor (Ketoprofen 10% Cream) Compared With Placebo in the Treatment of Acute Pain (Flare) Associated With Osteoarthritis of the Knee
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Imprimis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPI-110-002
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Acute Pain (Flare) Associated With Osteoarthritis (OA) of the Knee
MeSH Terms: conditions — Acute Pain | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Impracor (Ketoprofen 10% Cream) (Experimental): Topical Cream over a period of 14 days
  Interventions: Drug: Ketoprofen 10% Cream
- Placebo Cream: (Placebo Comparator): Topical Cream over a period of 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketoprofen 10% Cream
  Other Names: Impracor; IPI-110
  Arms: Impracor (Ketoprofen 10% Cream)
Drug: Placebo
  Arms: Placebo Cream:

SUMMARY:
The primary objective of the study is to assess analgesic efficacy of Impracor (Ketoprofen 10% Cream) compared to placebo for acute pain associated with OA flare of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of OA of the knee according to the ACR criteria.
* Kellgren-Lawrence grade 2-3 disease
* Be willing to stop taking all analgesics including NSAIDs and opioids for the duration of the study, with exception of study-specified rescue medication.

Exclusion Criteria:

* Total knee replacement surgery tentatively scheduled within next 6 months.
* Palpable knee effusion.
* Significant pain outside the target knee, including significant hip, back, or contralateral knee pain.
* Any type of orthopedic and/or prosthetic device or any skin abnormalities on the target knee that would prevent evaluations of local tolerability.
* History of asthma, rheumatoid arthritis, chronic inflammatory disease (e.g., colitis), or fibromyalgia.
* History of gastrointestinal bleeding or peptic ulcer disease within the past 3 years.
* Have a positive urine drug test for illegal drug substances, non-prescribed controlled substances, or alcohol at screening.
* Acute or chronic illness that in the opinion of the investigator could compromise the integrity of study data or place the subject at risk by participating in the study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be measured by changes in WOMAC pain subscale scores calculated by comparing baseline WOMAC pain subscale scores on Day 1 to the average WOMAC Pain Subscale scores on Day 4, 6, and 8. | Day 4, 6 and 8

SECONDARY OUTCOMES:
Change in Patient Global Assessment of knee arthritis using the modified Patient Overall Health Assessment from Day 1 to Day 8. | Day 8